CLINICAL TRIAL: NCT03208608
Title: The Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals (RBANS-H) in Older Adults With Normal Hearing or Age-related Hearing Loss
Brief Title: The RBANS-H in Older Adults With Normal Hearing or Age-related Hearing Loss
Acronym: RBANS-H_ARHL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZA, Principal investigator, University Hospital, Antwerp
Other Study IDs: 16/43/450
Record Dates: First submitted 2017-06-23; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Normal Hearing
Keywords: RBANS-H; Older adults; Normal hearing; Cognition; Age-related hearing loss
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Normal hearing older adults: Older adults with normal hearing or age-related hearing loss
  Interventions: Diagnostic Test: RBANS-H

INTERVENTIONS:
Diagnostic Test: RBANS-H — The RBANS-H is a diagnostic cognitive test battery

SUMMARY:
The present cross-sectional study aims to examine the cognitive capabilities of older adults, aged 50 to 89, with normal hearing or age-related hearing loss by means of the Repeatable Battery for the Assessment of Neuropsychological Status for Hearing impaired individuals (RBANS-H). Secondly, the correlations between cognition on the one hand and hearing and speech reception capabilities on the other hand are investigated. For this purpose, twenty participants are included in the age categories 50 to 59, 60 to 69, 70 to 79 and 80 to 89, bringing the total number to 80. Three questionnaires are administered to the participants: the Health Utilities Index-2/3 (HUI 2/3), Dizziness Handicap Inventory (DHI) and a general questionnaire on education and profession, medical history, hearing aid use and tinnitus. Also an audiological examination is performed, including pure tone audiometry, speech in quiet and speech in noise audiometry. Finally, cognition is assessed using the RBANS-H.

ELIGIBILITY:
Inclusion Criteria:

* Hearing: Air conduction hearing thresholds according to age, based on the ISO standards
* Age: 50 - 89

Exclusion Criteria:

* History of any neurological disease
* History of otological surgery or disease

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 to 89 with hearing thresholds according to their age and without history of any neurological or otological diseases
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
RBANS-H total scaled score | Baseline
  The RBANS-H assess cognition and provides one total score of cognition.

SECONDARY OUTCOMES:
RBANS-H index scores | Baseline
  The RBANS-H assesses five cognitive domains (Immediate Memory, Visuospatial/constructional, Language, Attention and Delayed Memory). The test consists of twelve subtests and the score on each subtest contributes to one of the five domains.
Free field best aided speech in noise audiometry: Speech Reception Threshold (SRT) | Baseline
  The speech reception in noise is assessed by means of the Leuven Intelligibility Sentences Test (LIST) using an adaptive procedure. This speech material is developed to quantify the speech understanding in subjects with severely impaired hearing. The frequency spectrum of the noise signal is equal to the long-term average speech spectrum of the sentences. The level of the noise is fixed at 65 dB SPL, while the level of the speech signal is altered depending on the response of the patient. Each list consists of ten sentences and the speech reception threshold (SRT) is calculated as the mean level of the last five sentences together with the level of the imaginary 11th sentence of the list. This speech in noise test is performed both pre- and postoperatively in an aided, free field situation with the loudspeaker in front of the subject at a distance of one meter.
Free field best aided speech in quiet audiometry (phoneme score): SRT | Baseline
  Speech reception in quiet is measured using Dutch open-set word lists. Each list consists of twelve monosyllabic words (consonant-vowel-consonant) of which one is a training item. The lists are presented at 65, 55, 40, 30, 20 and 10 dB SPL in free field with a loudspeaker at 0° azimuth. The intensity at which 50% of the phonemes is received correctly, is the SRT.
Free field best aided hearing thresholds: Fletcher Index (FI) | Baseline
  The best aided thresholds with no, one or two hearing aid(s) are measured through free field audiometry with warble tones. The loudspeaker is placed at a distance of one meter in front of the subject at ear level.
Health Utilities Index-2/3 (HUI 2/3) | Baseline
  The HUI questionnaire measures the self-perceived health status of the participant and rates the health-related quality of life (HRQL). The questionnaire consists of 17 items with four to six options. The HRQL scoring systems provide utility (preference) scores on a generic scale where dead = 0.00 and perfect health = 1.00.
Dizziness Handicap Inventory (DHI) | Baseline
  The DHI is used to quantify the impact of dizziness on everyday life. This 25-item questionnaire was developed to assess the self-perceived handicapping effects imposed by vestibular system disorders. Each item is rated as Yes = 4, Sometimes = 2 or No = 0 and contributes to one of three subscales, namely Functional, Emotional and Physical. A total score is calculated adding the scores on each item.
General questionnaire | Baseline
  A non-validated general questionnaire on education and profession, medical history, hearing aid use and tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Paul Van de Heyning, prof PhD MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium